CLINICAL TRIAL: NCT04650009
Title: Physical Activity in Children With Inherited Cardiac Diseases : a Qualitative
Brief Title: Physical Activity in Children With Inherited Cardiac Diseases
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Paediatric Cardiology and Rehabilitation Unit, St-Pierre Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0118
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Long QT Syndrome; Brugada Syndrome; Catecholaminergic Polymorphic Ventricular Tachycardia; Hypertrophic Cardiomyopathy; Dilated Cardiomyopathy
Keywords: Arrythmogenic right ventricular cardiomyopathy; Physical activity; Inherited cardiac disease; Peadiarics
MeSH Terms: conditions — Long QT Syndrome; Brugada Syndrome; Polymorphic Catecholaminergic Ventricular Tachycardia; Cardiomyopathy, Hypertrophic; Cardiomyopathy, Dilated; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Use lay language.

Current guidelines regarding physical activity in patients with inherited arrhythmia and cardiomyopathy are mostly dedicated to adult patients, with a special focus on sports competition. Their application to the pediatric population has been scarcely evaluated.

Physical activity is well known for its health benefits but may be dangerous in this population, which leads to confusion within the medical community and among patients. Actual physical activity of children with such inherited cardiac disorders is unknown.

This study aimed to assess the level of physical activity in children with inherited arrhythmia and cardiomyopathy, and the adherence to the current European guidelines on the subject. Secondary objectives aimed to assess through a qualitative analysis the impact of the disease on physical activity and daily life in this population.

The level of physical activity and adherence to current guidelines will be determined from interviews between the patient and the principal investigator. Each patient will be questioned in order to explore the experiences, motivations and feelings of participants regarding physical activity. The standardized questionnaire was created by the principal investigator and members of the clinical research team.

The investigators believe that many children practice physical activity outside the current guidelines and hope to identify the main determinants of physical activity in this population.

ELIGIBILITY:
Inclusion criteria:

Children from 6 to 18 years old with clinical and/or genetic diagnosis of :

* Long QT syndrome
* Brugada syndrome
* Catecholaminergic polymorphic ventricular tachycardia
* Hypertrophic cardiomyopathy
* Dilated cardiomyopathy
* Arrythmogenic right ventricular cardiomyopathy

Exclusion criteria:

* Presence of extra cardiac co-morbidity with motor or psychological repercussions hingering physical activity
* Refusal from children or parent to participate in the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will take place in two paediatric tertiaty hospitals : the paediatric and congenital cardiology department of Montpellier university hospital and the paediatric cardiology and rehabilitation unit of St-Pierre institute in Palavas-Les-Flots, France.
  Children aged from 6 to 18 years old with genetic and/or clinical diagnosis of inherited cardiomyopathies (hypertrophic cardiomyopathy, dilated cardiomyopathy and arrythmogenic right ventricular cardiomyopathy) or inherited primary arrhythmia syndrome (long QT syndrome, brugada syndrome and catecholaminergic polymorphic ventricular tachycardia) are eligible to participate in this study. Each subject accepting to participate during the annual follow up consultation will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Proportion of children with inheritec cardiac disorders respecting the current European guidelines on sports cardiology and exercise (ESC 2020). | 1 day
  Patient's physical activity will be analysed to evaluate the adherence to current European guidelines regarding physical activity. Patients will be categorized into 3 groups, upon the level of adherence to the guidelines (complete adherence, partial adherence et no adherence).

SECONDARY OUTCOMES:
Qualitative analysis evaluating the psychological and emotional impact of physical activity restriction on daily life. | 1 day
  Patients will be interviewed by the principal investigator for 20 to 30 minutes with a focus on physical activity, in order to collect motivations, feelings and discourse of the patient, classified in main themes (positive, negative or neutral).
  No score is used in this study:
  The secondary outcome is a qualitative analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD-PhD, Study Director — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Background] Boisson A, De La Villeon G, Huguet H, Abassi H, Pasquie JL, Lavastre K, Matecki S, Guillaumont S, Requirand A, Calderon J, Amedro P. Physical activity and aerobic fitness in children with inherited cardiac diseases. Arch Cardiovasc Dis. 2021 Nov;114(11):727-736. doi: 10.1016/j.acvd.2021.07.004. Epub 2021 Oct 27. PMID 34756533